CLINICAL TRIAL: NCT01141387
Title: Clinical Outcomes in MEasurement-Based Treatment (COMET)
Brief Title: Outcomes in MEasurement-Based Treatment
Acronym: COMET
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Study Director, Bristol -Myers Squibb
Other Study IDs: CN138-534
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2011-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients at the intervention sites: The intervention sites will receive the results of the patient-reported depression severity collected during the phone interviews on a monthly basis. The patients in the intervention arm will be interviewed by phone once per month for 6 months.
- Patients at the usual care sites: The usual care sites will receive the results of the patient-reported depression severity at the end of the study. Patients in the usual care arm will be interviewed at 3 months and 6 months post study enrollment.

SUMMARY:
The primary objective for this study is to assess the impact of a measurement based treatment program (MBT) on Major Depressive Disorder (MDD) remission rates in patients whose primary care provider (PCP) receives monthly patient-reported depression severity reports compared to patients whose PCP does not receive monthly reports.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Diagnosis of major depressive disorder
* Prescribed a new prescription for an antidepressant medication on the date of study enrollment and currently taking the medication 'New' is defined as no antidepressant use in the previous 120 days
* Primary depression management is performed by the primary care provider
* Capable of self-management (i.e., taking medications and independently responding to follow-up contacts)
* Able to provide informed consent to participate
* Sufficient ability as judged by the physician to read, understand and complete survey instruments written in English and phone interviews spoken in English

Exclusion Criteria:

* History psychotic disorder or bipolar disorder
* Diagnosis of current postpartum depression
* Diagnosis of bereavement less than 8 weeks duration
* Currently pregnant
* History of suicide attempts or current suicide plan
* Need for psychiatric hospitalization at enrollment visit
* History of adjunctive treatments including electroconvulsive treatment (ECT), vagus nerve stimulation (VNS), transcranial magnetic stimulation (TMS), magnetic seizure therapy (MST), or deep brain stimulation (DBS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 914 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Remission rate assessed by the Patient Health Questionnaire - 9 item (PHQ-9) instrument | Measured at baseline
Remission rate assessed by the Patient Health Questionnaire - 9 item (PHQ-9) instrument | Follow-up upto 6 months

SECONDARY OUTCOMES:
Response rate assessed by the PHQ-9 instrument | 6 months
The medication prescribed including refills, dose titrations, switching and augmentation | 6 months
Health care utilizations including office visits, emergency room visits and hospitalization | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm